CLINICAL TRIAL: NCT06916143
Title: A Phase 1, Open-label, Randomized, Four-way Crossover Study to Assess the Relative Bioavailability of Two Phase 3 LY4100511 (DC-853) Tablet Formulations Compared With the Phase 2 LY4100511(DC-853) Tablet Formulation, With and Without a Proton Pump Inhibitor in Healthy Participants
Brief Title: Comparing the Extent to Which Three Different Formulations of LY4100511 (DC-853) Are Made Available in the Body, Alone and in the Presence of a Drug That Reduces Stomach Acid
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27274; J5C-MC-FOAH, DCE853105 (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY4100511 (DC-853) + Rabeprazole - Reference (Experimental): LY4100511 (DC-853) administered orally alone then LY4100511 (DC-853) administered orally with Rabeprazole.
  Interventions: Drug: LY4100511; Drug: Rabeprazole
- LY4100511 (DC-853) + Rabeprazole - Test 1 (Experimental): LY4100511 (DC-853) administered orally alone and then LY4100511 (DC-853) administered orally with Rabeprazole.
  Interventions: Drug: LY4100511; Drug: Rabeprazole
- LY4100511 (DC-853) + Rabeprazole - Test 2 (Experimental): LY4100511 (DC-853) administered orally alone and then LY4100511 (DC-853) administered orally with Rabeprazole
  Interventions: Drug: LY4100511; Drug: Rabeprazole

INTERVENTIONS:
Drug: LY4100511 — Administered orally.
Drug: Rabeprazole — Administered orally.

SUMMARY:
The main purpose of this study is to compare the bioavailability of 3 different formulations of LY4100511 and if the use of a proton pump inhibitor (PPI) alters the bioavailability of the 3 different formulations.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kilograms per meter squared (kg/m2), inclusive, and a body weight of ≥50 kg.
* In good health, as determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG) and vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in, and from the physical examination at check-in, as assessed by the Investigator (or designee).

Exclusion Criteria:

* Have a 12-lead ECG abnormality that, in the opinion of the Investigator,

  * increases the risk associated with participating in the study
  * may confound ECG data analysis
  * a QTcF: >450 millisecond (msec) for males, or >470 msec for females
  * short PR interval <120 msec or PR interval >220 msec
  * second or third degree atrioventricular block
  * intraventricular conduction delay with QRS >120 msec
  * complete right bundle branch block
  * left bundle branch block, or
  * Wolff Parkinson-White syndrome
* Have a current or recent acute, active infection (for example, for a least 30 days before screening and up to Day -1, participants must have no symptoms or signs of infection in the absence of any anti-infective treatment).
* Had any malignancy within the past 5 years. Exceptions: successfully treated basal cell skin carcinoma or squamous cell skin carcinoma, with no evidence of recurrence or metastatic disease within the 3 years prior to baseline.
* Have inflammatory bowel disease (IBD), including ulcerative colitis or Crohn's disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK): Area Under the Concentration Curve from 0 to Infinity (AUC0-∞) of LY4100511 (DC-853) | Predose up to 26 Days
  PK: AUC0-∞ of LY4100511
Pharmacokinetic (PK): Maximum Concentration (Cmax) of LY4100511 (DC-853) | Predose up to 26 Days
  PK: Cmax of LY4100511 (DC-853)
Pharmacokinetic (PK): Area Under the Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-T) of LY4100511 (DC-853) | Predose up to 26 Days
  PK: AUC0-T of LY4100511 (DC-853)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No